CLINICAL TRIAL: NCT04184596
Title: Preferences in Pain Treatment: A Discrete Choice Experiment in Patients With Peripheral Neuropathic Pain (pNP)
Acronym: DExPri
Status: Completed | Type: Observational
Sponsor: LinkCare GmbH (Industry)
Collaborators: Schmerzpraxis Wiesbaden (Unknown); Schmerz- und Palliativzentrum Rhein-Main Wiesbaden (Unknown); Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: VF/1014/1070
Record Dates: First submitted 2019-11-29; First posted 2019-12-03 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Neuralgia Peripheral; Neuropathic Pain; Patient Preference
Keywords: Discrete Choice Experiment
MeSH Terms: conditions — Neuralgia; Patient Preference

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stated-Preferences Observational Group: A discrete choice experiment will be conducted with participants with peripheral neuropathic pain in the stated-preferences observational group. The instrument will measure patient preferences for topical versus systemic pain treatment.
  Interventions: Other: Discrete Choice Experiment

INTERVENTIONS:
Other: Discrete Choice Experiment — An online-based Discrete-Choice Experiment (DCE) using a survey for stated treatment preferences and socio-demographics. Furthermore, the neuropathic pain component will be assessed in all patients with the Numeric Pain Rating Scale instrument.

SUMMARY:
The objective of this study is to identify and weight attributes of topic and systemic pain treatment options relevant from the patients' perspective with peripheral neuropathic pain. The study will use a discrete choice experimental design to reach its objective.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed peripheral neuropathic pain (pNP) as assessed by study sites

Exclusion Criteria:

* Patients with no sufficient knowledge in written or oral German as assessed by study sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 150 patients will be included in this study. Participating centers are outpatient centers, specialist in pain treatment in the state of Hesse.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Patient preferences for topical and systemic pain treatment attributes | 20 minutes after survey start
  Utility values obtained via multinominal logit estimates from discrete choice experiment

SECONDARY OUTCOMES:
Relevance of attributes attributed with topical and systemic pain treatment | 5 minutes after survey start
  Derived from Likert scale
Marginal rate of substitution against pain reduction | 20 minutes after survey start
  Derived from discrete choice experiment

CONTACTS AND LOCATIONS:
Overall Officials: Tino Schubert, MSc, Study Chair — LinkCare GmbH
Locations (3):
- Germany (3):
  - LinkCare GmbH, Stuttgart, Baden-Wurttemberg
  - Schmerz- und Palliativzentrum Rhein-Main, Wiesbaden, Hesse
  - Schmerzpraxis Wiesbaden, Wiesbaden, Hesse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schubert T, Kern KU, Schneider S, Baron R. Oral or Topical Pain Therapy-How Would Patients Decide? A Discrete Choice Experiment in Patients with Peripheral Neuropathic Pain. Pain Pract. 2021 Jun;21(5):536-546. doi: 10.1111/papr.12989. Epub 2021 Feb 1. PMID 33342078